CLINICAL TRIAL: NCT04924439
Title: Effects Reflexology on Postpartum Pain, Fatigue, Sleep Quality and Lactation
Brief Title: Effects of Reflexology on Postpartum Pain, Fatigue, Sleep Quality and Lactation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Gaziantep (Other)
Responsible Party: Principal Investigator, Aysegul Kilicli, Nursing, University of Gaziantep
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: reflexology and cesarean
Record Dates: First submitted 2021-06-03; First posted 2021-06-14 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Breast Feeding; Fatigue; Sleep; Pain, Postoperative
Keywords: fatigue; lactation; pain; postpartum; sleep quality; reflexology
MeSH Terms: conditions — Breast Feeding; Fatigue; Pain, Postoperative; Pain; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Small papers with 40 experiments and 40 controls were folded and put into closed, sealed, opaque envelopes, then all the envelopes were put in a bag and mixed. The women were asked to choose one envelope from the bag, and it was determined whether the experimental or control group they were included in before the application. The women in the study did not know which of the experimental and control groups they were included in, and the statistical analysis was planned double-blind, as an independent statistician apart from the researchers did it.
  Statistical analysis of the research was carried out independently by a statistician.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (foot reflexology group) (Experimental): Primiparas appropriate for the criteria, admitted to the clinic due to CS and accepting to participate in the study were randomly placed into groups. Reflexology was performed in the intervention group mothers, and the questionnaires and scales were self-reportingly filled in by the lead researcher (SC).
  Different rooms were allocated for the participants in the intervention and control groups not to affect each other.
  Foot reflexology was applied to the experimental group for 40 minutes once a week for postpartum 8 weeks.
  Interventions: Other: foot reflexology
- control group (No Intervention): Primiparas appropriate for the criteria, admitted to the clinic due to CS and accepting to participate in the study were randomly placed into groups. Reflexology was performed in the intervention group mothers, and the questionnaires and scales were self-reportingly filled in by the lead researcher (SC).
  Different rooms were allocated for the participants in the intervention and control groups not to affect each other.

INTERVENTIONS:
Other: foot reflexology — Foot reflexology was applied to the experimental group for 40 minutes once a week for postpartum 8 weeks. The control group was only watched.
  Arms: experimental group (foot reflexology group)

SUMMARY:
The aim of this research is to determine the effect of foot reflexology applied to primiparous women who had cesarean section in the postpartum period on pain, fatigue, sleep quality and lactation. This research is a randomized controlled trial. The study was conducted in Şanlıurfa, which has the highest fertility rate in Turkey.

DETAILED DESCRIPTION:
The aim of this research is to determine the effect of foot reflexology applied to primiparous women who had cesarean section in the postpartum period on pain, fatigue, sleep quality and lactation. This research is a randomized controlled trial. The study was conducted in Şanlıurfa, which has the highest fertility rate in Turkey. The sample of the research consisted of 80 primiparous women (reflexology group: 40 and control group: 40). The data were collected between 01 January 2020 - 31 January 2021. "Introductory Information Form", "Visual Analogue Scale" for Pain, "Visual Analog Scale for Fatigue", "Pittsburg Sleep Quality Index" and "Bristol Breastfeeding Assessment Tool" were used as data collection tools. Foot reflexology was applied to the experimental group for 40 minutes (left foot 20 minutes and right foot 20 minutes) once a week for postpartum 8 weeks. The control group was only watched. In the intergroup comparison of the experimental and control groups, chi-square for categorical variables and independent groups t-test for numerical variables were used. Two-way repeated measures ANOVA test was performed in terms of time and group interaction in repeated measurements

ELIGIBILITY:
Inclusion Criteria:

* Caesarean section,
* Primipary,
* 19 and over and under 35
* Literate,
* 37 and above pregnancy week
* Giving birth singularly,
* Having spinal anesthesia
* No chronic disease or pregnancy complication,
* Have no breast-related health problems
* Have not had an operation related to the breast,
* Women who do not have any health problems in the feet of the mothers in the treatment group

Exclusion Criteria:

* The baby has died or is not present,
* Multiparous,
* Women with health problems in their feet

Ages: 19 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | Change from Visual Analogue Scale (VAS) scores at first, second, third, fourth, fifth, sixth, seventh and eighth week after cesarean. ]
  The scale developed by Huskisson (1974) is used for pain assessment in musculoskeletal system and other clinical assessments. VAS is used to convert some values that cannot be measured numerically to numeric. It is a frequently used measurement tool because it is easy and safe to apply. The words "I have no pain" on the left end of the 10 cm long horizontal line and "I have pain" on the right end. The individual is asked to mark the point on this horizontal line that best expresses the severity of pain in his body. The distance from the point marked by the individual to the left end is measured and the pain score is determined. It is evaluated that the severity of the pain increases as the VAS value approaches 10, and decreases as it approaches 0. The lowest 0 and the highest 10 points are taken from the scale.
Visual Similarity Scale for Fatigue (YSSF) | Change from Visual Similarity Scale for Fatigue (YSSF) scores at first, second, third, fourth, fifth, sixth, seventh and eighth week after cesarean. ]
  It is in the form of a 10 cm ruler with the most positive statements on one end of the scale and the most negative statements on the other. The most positive expression of the fatigue sub-dimension is 0, the most negative expression is 10, the most negative expression of the energy sub-dimension is 0, and the most positive expression is 10. A high score of the fatigue sub-dimension and a low score of the energy sub-dimension indicate a high severity of fatigue. The calculation method of the scale is determined by adding up all the scores obtained from the scale items. The lowest score for YSSF is 0, and the highest score is 180. The lowest score for the YSSF fatigue sub-dimension is 0, and the highest score is 130. The lowest score is 0 for the energy sub-dimension of YSSF and the highest score is 50. The scale does not have a cut-off point.
Pittsburg Sleep Quality Index (PSQI) | Change from Pittsburg Sleep Quality Index (PSQI) scores at first, fourth and eighth week after cesarean. ]
  In order to evaluate the sleep quality in the last month, Buysse et al. (1989) is a quantitative measure of sleep quality as good and bad sleep. Its Turkish adaptation was done by Ağargün et al. (1996), Cronbach's α internal consistency coefficient is 0.80. It consists of a total of 24 questions and 7 sub-components. 18 items and 7 sub-components are included in the scoring. Each item is evaluated as 0-3 points and the sum of 7 sub-components forms the PSQI score. The lowest score of the scale is 0 and the highest score is 21. A total PSQI score of ≤5 indicates good sleep, and >5 indicates poor sleep.
Bristol Breastfeeding Assessment Tool (BBAT) | Change from Bristol Breastfeeding Assessment Tool (BBAT) scores at first, second, third, fourth, fifth, sixth, seventh and eighth week after cesarean. ]
  Each item in the scoring of the scale is between 0-2 points. The calculation method is the sum of all scores obtained from the scale items. The lowest score obtained from the scale is 0, and the highest score is 8. The scale does not have a breakpoint. A low score indicates that breastfeeding is ineffective, and a high score indicates that breastfeeding is effective.

CONTACTS AND LOCATIONS:
Overall Officials: simge zeyneloğlu, proffessor, Study Director — GAZİANTEP UNİVERSİTY CLINICAL RESEARCH ETHICS COMMITTE
Locations (1):
- Gaziantep University Health Sciences Enstitutes, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No